CLINICAL TRIAL: NCT06174129
Title: Prevalence and Factors Associated With Atrial Fibrillation in Patients With Type 2 Diabetes: A Case-Control Study
Brief Title: Prevalence and Factors Associated With Atrial Fibrillation in Patients With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Burapha University (Other)
Responsible Party: Principal Investigator, Sukrisd Koowattanatianchai, Assistant Professor Dr., Burapha University
Other Study IDs: HS114/2565
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Atrial Fibrillation; Type 2 Diabetes
MeSH Terms: conditions — Atrial Fibrillation; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Type 2 diabetes patients with atrial fibrillation: The 12-lead electrocardiography recordings of type 2 diabetes patients were reviewed by a cardiologist to confirm the presence of atrial fibrillation. The clinical parameters, including age, sex, body-mass index, underlying medical conditions, blood pressure, heart rate, type 2 diabetes duration, laboratory values, and medications were analyzed and compared between atrial fibrillation and non-atrial fibrillation patients.
  Interventions: Other: Routine examinations
- Type 2 diabetes patients without atrial fibrillation: The 12-lead electrocardiography recordings of type 2 diabetes patients were reviewed by a cardiologist to confirm the presence of atrial fibrillation. The clinical parameters, including age, sex, body-mass index, underlying medical conditions, blood pressure, heart rate, type 2 diabetes duration, laboratory values, and medications were analyzed and compared between atrial fibrillation and non-atrial fibrillation patients.
  Interventions: Other: Routine examinations

INTERVENTIONS:
Other: Routine examinations — Electrocardiography and clinical parameters examinations, including age, sex, body-mass index, underlying medical conditions, blood pressure, heart rate, type 2 diabetes duration, laboratory values, and medications

SUMMARY:
This case-control study was conducted at Burapha University Hospital. The 12-lead electrocardiography recordings of type 2 diabetes patients were reviewed by a cardiologist to confirm the presence of atrial fibrillation. The clinical parameters, including age, sex, body-mass index, underlying medical conditions, blood pressure, heart rate, type 2 diabetes duration, laboratory values, and medications were analyzed and compared between atrial fibrillation and non-atrial fibrillation patients.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with type 2 diabetes who visited the medical clinic between June 2022 and June 2023

Exclusion Criteria:

* Patients with missing information on the urinary albumin value and electrocardiograms at the latest date

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Outpatients with type 2 diabetes who visited the medical clinic at Burapha University Hospital, Chonburi province, Thailand between June 2022 and June 2023 were enrolled in the present study.
Sampling Method: Non-Probability Sample
Enrollment: 427 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of atrial fibrillation | June 2022 and June 2023
  Prevalence of atrial fibrillation in patients with type 2 diabetes
Factors associated with atrial fibrillation | June 2022 and June 2023
  Factors associated with atrial fibrillation in patients with type 2 diabetes, including age, hypertension, heart failure, thyroid disease, type 2 diabetes duration, body mass index, estimated glomerular filtration rate, glycated hemoglobin, presence of albuminuria, and use of diuretic medications

CONTACTS AND LOCATIONS:
Locations (1):
- Burapha University Hospital, Mueang, Changwat Chon Buri, Thailand

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.